CLINICAL TRIAL: NCT02163824
Title: A Phase III, Double-Masked, Randomized, Controlled Trial of KPI-121 in Postsurgical Inflammation
Brief Title: Safety and Efficacy of KPI-121 in Subjects With Postsurgical Inflammation
Acronym: Hawaii-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kala Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPI-121-C-001
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Ocular Infections, Irritations and Inflammations
Keywords: postsurgical; postoperative; ocular; cataract; inflammation; pain; corticosteroid
MeSH Terms: conditions — Eye Infections; Inflammation; Cataract; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- KPI-121 0.25% QID (Active Comparator): KPI-121 0.25% Ophthalmic Suspension dosed 4 times daily for 14 days after routine, uncomplicated surgery for cataract removal and intraocular lens implant.
  Interventions: Drug: KPI-121 0.25%
- KPI-121 1.0% BID (Active Comparator): KPI-121 1.0% Ophthalmic Suspension dosed 2 times daily for 14 days after routine, uncomplicated surgery for cataract removal and intraocular lens implant.
  Interventions: Drug: KPI-121 1.0%
- Vehicle of KPI-121 0.25% (Placebo Comparator): Vehicle of KPI-121 0.25% Ophthalmic Suspension dosed 4 times daily for 14 days after routine, uncomplicated surgery for cataract removal and intraocular lens implant.
  Interventions: Drug: Vehicle of KPI-121 0.25%
- Vehicle of KPI-121 1.0% (Placebo Comparator): Vehicle of KPI-121 1.0% Ophthalmic Suspension dosed 2 times daily for 14 days after routine, uncomplicated surgery for cataract removal and intraocular lens implant.
  Interventions: Drug: Vehicle of KPI-121 1.0%

INTERVENTIONS:
Drug: KPI-121 0.25% — KPI-121 drug product will be supplied as 0.25% as a suspension in identically packaged opaque dropper bottles. KPI-121 drug product is a sterile, aqueous, submicron suspension of loteprednol etabonate.
  Other Names: KPI-121 0.25% Ophthalmic Suspension; Loteprednol etabonate 0.25%
  Arms: KPI-121 0.25% QID
Drug: KPI-121 1.0% — KPI-121 drug product will be supplied as 1.0% as a suspension in identically packaged opaque dropper bottles. KPI-121 drug product is a sterile, aqueous, submicron suspension of loteprednol etabonate.
  Other Names: KPI-121 1.0% Ophthalmic Suspension; Loteprednol etabonate 1.0%
  Arms: KPI-121 1.0% BID
Drug: Vehicle of KPI-121 0.25% — Placebo control arms will receive the same bottles containing vehicle of KPI-121 including all components at the concentrations used in the KPI-121 drug product with the exception of the active component, loteprednol etabonate.
  Other Names: Vehicle of KPI-121 0.25% Ophthalmic Suspension
  Arms: Vehicle of KPI-121 0.25%
Drug: Vehicle of KPI-121 1.0% — Placebo control arms will receive the same bottles containing vehicle of KPI-121 including all components at the concentrations used in the KPI-121 drug product with the exception of the active component, loteprednol etabonate.
  Other Names: Vehicle of KPI-121 1.0% Ophthalmic Suspension
  Arms: Vehicle of KPI-121 1.0%

SUMMARY:
The primary purpose of this study is to determine the efficacy and safety of KPI-121 ophthalmic suspension compared to placebo in subjects who have undergone cataract surgery. The efficacy and safety of two different concentrations and two different dosing regimens of KPI-121 are also being assessed.

DETAILED DESCRIPTION:
This is a Phase III, multicenter, double-masked, randomized, placebo-controlled, parallel-group study designed to evaluate the efficacy and safety of two doses and two dosing regimens of KPI-121 ophthalmic suspension versus placebo in subjects who require treatment of postoperative anterior ocular inflammation.

Approximately 500 subjects will be screened and up to 402 subjects with one study eye each will be randomized in this study at approximately 25 centers located in the United States. Subjects who experience postoperative inflammation on the first day following routine, uncomplicated, cataract surgery and who meet all other eligibility criteria will be randomized to one of four study groups (0.25% four times daily or 1.0% two times daily) or Placebo A four times daily or Placebo B two times daily. Drug product or placebo will be initiated on the day following surgery and instilled as one to two drops in the study eye according to the assigned dosing regimen for 14 days.

This study will include up to 7 clinic visits (including the surgery day) over 18 to 33 days total study duration. Visit 1 (Screening) will occur between 14 to 1 day(s) prior to surgery, and subjects who meet preoperative screening inclusion/exclusion criteria will be entered into the study. At Visit 2 (Surgery/Day 0) subjects will undergo routine cataract surgery according to the Investigator's normal procedures. Visit 3 (Randomization/Day 1) will occur on the day following surgery.

Following randomization, subjects will be instructed to return to the clinic to be evaluated at Visit 4 (Day 3 +2 day), Visit 5 (Day 8 ±1 day), and Visit 6 (Day 15 ±1 day). The last dose of study product will be administered upon completion of 14 days of evaluation. Following the End of Study Product Use Visit (Visit 6; Day 15 ±1 day), subjects will be asked to return to the clinic on Day 17-19 for Visit 7 (Follow-Up) and will be released from the study.

ELIGIBILITY:
FURTHER STUDY DETAILS PROVIDED BY KALA PHARMACEUTICALS, INC.

Inclusion Criteria:

* Candidates for routine, uncomplicated cataract surgery
* In Investigator's opinion, potential postoperative Snellen Distance VA by pinhole method of at least 20/200 in study eye.

Exclusion Criteria:

* Known hypersensitivity/contraindication to study product(s) or components.
* History of glaucoma, IOP >21 mmHg at the screening or randomization visits, or being treated for glaucoma in either eye.
* Diagnosis of: ongoing ocular infection; severe/serious ocular condition that in judgment of Investigator could confound study assessments or limit compliance; severe/serious systemic disease or uncontrolled medical condition that in judgment of Investigator could confound study assessments or limit compliance; or have been exposed to an investigational drug within the 30 days prior to screening or 19 days following surgery.
* In the opinion of Investigator or study coordinator, be unwilling or unable to comply with study protocol or unable to successfully instill eye drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Sall Research Medical Center, Artesia, California
  - North Valley Eye Medical Group, Mission Hills, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Clayton Eye Center, Morrow, Georgia
  - Price Vision Group, Indianapolis, Indiana
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Taustine Eye Center, Louisville, Kentucky
  - Tauber Eye Center, Kansas City, Missouri
  - Tekwani Vision Center, St Louis, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Ophthalmology Consultants, St Louis, Missouri
  - Las Vegas Physicians Research Group, Henderson, Nevada
  - Raymond Fong, MDPC, New York, New York
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - Cornerstone Eye Care, High Point, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - The Eye Center of Columbus, Columbus, Ohio
  - Westside Research, LLC, Spartanburg, South Carolina
  - The Eye Clinic of Texas, Affiliate of Houston Eye Associates, League City, Texas
  - R&R Eye Research, LLC, San Antonio, Texas
  - Kozlovsky Delay & Winter Eye Consultants, LLC, San Antonio, Texas
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle of KPI-121: Vehicle of KPI-121 0.25% Ophthalmic Suspension dosed 4 times daily or 1.0% Ophthalmic Suspension dose 2 times daily for 14 days after routine, uncomplicated surgery for cataract removal and intraocular lens implant.
  Vehicle of KPI-121: Placebo control arms will receive the same bottles containing vehicle of KPI-121 including all components at the concentrations used in the KPI-121 drug product with the exception of the active component, loteprednol etabonate.
Period: Overall Study
Arm/Group | KPI-121 0.25% QID | KPI-121 1.0% BID | Vehicle of KPI-121
Started | 129 | 125 | 126
Completed | 127 | 124 | 124
Not Completed | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KPI-121 0.25% QID | KPI-121 1.0% BID | Vehicle of KPI-121 | Total
Number analyzed (Participants) | 129 | 125 | 126 | 380
Age, Continuous [Mean (Full Range); unit: years] | 68.4 [34 to 88] | 67.9 [41 to 89] | 69.8 [52 to 87] | 68.7 [34 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 75 | 78 | 226
  Male | 56 | 50 | 48 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 15 | 13 | 36
  Not Hispanic or Latino | 121 | 110 | 113 | 344
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 21 | 19 | 21 | 61
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 1 | 5
  Black or African American | 7 | 9 | 14 | 30
  White | 96 | 91 | 87 | 274
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 2 | 4 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 129 | 125 | 126 | 380

OUTCOME MEASURES:

1. Primary Outcome: Resolution of Anterior Chamber Cells
Description: Subjects with complete resolution of anterior chamber cells (cell score = 0) without rescue medication at Day 8/Visit 5 and Day 15/Visit 6.
  0= No cells seen
  1. 1 to 5 cells
  2. 6 to 15 cells
  3. 16 to 30 cells
  4. greater than 30 cells
Time Frame: Visit 5 (postoperative day 8) and Visit 6 (postoperative day 15)
Population: Intent to treat- all subjects randomized
Measure: Count of Participants; unit: Participants
Arm/Group | KPI-121 0.25% QID | KPI-121 1.0% BID | Vehicle of KPI-121
Number analyzed (Participants) | 129 | 125 | 126
Participants | 48 | 39 | 19
Statistical Analysis 1: Comparison: KPI-121 1.0% BID vs Vehicle of KPI-121; All statistical tests of hypotheses performed for the pairwise comparison of means were two-sided. All statistical tests employed a level of significance of alpha = 0.05; Test type: Superiority; p = .0024, Chi-squared; Difference in % of responders = 16.1, 95% CI 2-sided [5.9 to 26.4] — Estimated Value is the between-group difference for % of responders and is expressed as a percentage
Statistical Analysis 2: Comparison: KPI-121 0.25% QID vs Vehicle of KPI-121; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .0001, Chi-squared; Difference in % of responders = 22.1, 95% CI 2-sided [11.7 to 32.6] — Estimated Value is the between-group difference for % of responders and is expressed as a percentage

2. Primary Outcome: Resolution of Ocular Pain
Description: Subjects with complete resolution of pain (grade = 0) without rescue medication at Day 8/Visit 5 and Day 15/Visit 6.
Time Frame: Visit 5 (postoperative day 8) and Visit 6 (postoperative day 15)
Population: Intent to Treat- all subjects randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | KPI-121 0.25% QID | KPI-121 1.0% BID | Vehicle of KPI-121
Number analyzed (Participants) | 129 | 125 | 126
Participants | 73 | 67 | 43
Statistical Analysis 1: Comparison: KPI-121 1.0% BID vs Vehicle of KPI-121; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .0019, Chi-squared; Difference in % of responders = 19.5, 95% CI 2-sided [7.4 to 31.5] — Estimated Value is the between-group difference for % of responders and is expressed as a percentage
Statistical Analysis 2: Comparison: KPI-121 0.25% QID vs Vehicle of KPI-121; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .0003, Chi-squared; Difference in % of responders = 22.5, 95% CI 2-sided [10.6 to 34.4] — Estimated Value is the between-group difference for % of responders and is expressed as a percentage

3. Secondary Outcome: Anterior Chamber Cell Grade at Visit 5.
Description: Mean Grade of Anterior Chamber Cells (Scale 0-4) at Visit 5/Day 8. The difference in mean grade of AC cell count grade at Day 8 for KPI-121 1% dosed twice daily (BID) or 0.25% dosed four times daily (QID) compared with vehicle (either dosed BID or QID). Investigators were asked to grade AC cell based on the following scale wherein higher scores indicate a higher degree of cells present and a decrease across time indicates the condition is getting better.
  Anterior Chamber Cells 0 = No cells seen
  1. 1 - 5 cells
  2. 6 - 15 cells
  3. 16 - 30 cells 4 = greater than 30 cells
Time Frame: Visit 5 (postoperative day 8)
Population: Intent to Treat population minus subjects in each treatment group that discontinued the study by this time point or otherwise did not have this assessment completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% QID | KPI-121 1.0% BID | Vehicle of KPI-121
Number analyzed (Participants) | 128 | 125 | 125
score on a scale | 0.7 (0.73) | 0.9 (0.74) | 1.0 (0.86)
Statistical Analysis 1: Comparison: KPI-121 0.25% QID vs Vehicle of KPI-121; Test type: Superiority; p = 0.0007, ANCOVA; Mean Difference (Final Values) = -0.3 — Estimated value is the between-group difference in mean AC grade at Day 8
Statistical Analysis 2: Comparison: KPI-121 1.0% BID vs Vehicle of KPI-121; Test type: Superiority; p = 0.0440, ANCOVA; Mean Difference (Final Values) = -0.2 — Estimated value is the between-group difference in mean grade AC at Day 8

4. Secondary Outcome: Anterior Chamber Cell Grade at Visit 6.
Description: Mean Grade of Anterior Chamber Cells (Scale 0-4) at Visit 6/Day 15. The difference in mean grade of AC cell count grade at Day 15 for KPI-121 1% dosed twice daily (BID) or 0.25% dosed four times daily (QID) compared with vehicle (either dosed BID or QID). Investigators were asked to grade AC cell based on the following scale wherein higher scores indicate a higher degree of cells present and a decrease across time indicates the condition is getting better.
  Anterior Chamber Cells 0 = No cells seen
  1. 1 - 5 cells
  2. 6 - 15 cells
  3. 16 - 30 cells 4 = greater than 30 cells
Time Frame: Visit 6 (postoperative day 15)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% QID | KPI-121 1.0% BID | Vehicle of KPI-121
Number analyzed (Participants) | 127 | 124 | 124
score on a scale | 0.4 (.65) | 0.5 (.69) | 0.6 (.75)
Statistical Analysis 1: Comparison: KPI-121 0.25% QID vs Vehicle of KPI-121; Test type: Superiority; p = 0.0391, ANCOVA; Mean Difference (Final Values) = -0.2 — Estimated value is the between-group difference in mean AC grade at Day 15
Statistical Analysis 2: Comparison: KPI-121 1.0% BID vs Vehicle of KPI-121; Test type: Superiority; p = 0.1811, ANCOVA; Mean Difference (Final Values) = -0.1 — Estimated value is the between-group difference in mean AC grade at Day 15

5. Secondary Outcome: Ocular Pain Grades at Day 8.
Description: Mean Grade of Ocular Pain (Scale 0-5) at Visit 5/Day 8. The difference in mean grade of ocular pain grade at Day 8 for KPI-121 1% dosed twice daily (BID) or 0.25% dosed four times daily (QID) compared with vehicle (either dosed BID or QID). Subjects were given the Subject-Rated Ocular Pain Assessment to subjectively rate their pain. Higher scores were worse outcomes.
  The following scoring scale was used for ocular pain:
  0 = None
  1. Minimal
  2. Mild
  3. Moderate
  4. Moderately Severe
  5. Severe
Time Frame: Visit 5 (postoperative day 8)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% QID | KPI-121 1.0% BID | Vehicle of KPI-121
Number analyzed (Participants) | 128 | 125 | 125
score on a scale | 0.4 (0.74) | 0.4 (0.64) | 0.5 (0.89)
Statistical Analysis 1: Comparison: KPI-121 0.25% QID vs Vehicle of KPI-121; Test type: Superiority; p = 0.1953, ANCOVA; Mean Difference (Final Values) = -0.1 — Estimated value is the between-group difference in mean ocular pain grade at Day 8
Statistical Analysis 2: Comparison: KPI-121 1.0% BID vs Vehicle of KPI-121; Test type: Superiority; p = 0.0307, ANCOVA; Mean Difference (Final Values) = -0.2 — Estimated value is the between group difference of mean ocular pain grade at Day 8

6. Secondary Outcome: Ocular Pain Grades at Day 15.
Description: Mean Grade of Ocular Pain (Scale 0-5) at Visit 6/Day 15. The difference in mean grade of ocular pain grade at Day 15 for KPI-121 1% dosed twice daily (BID) or 0.25% dosed four times daily (QID) compared with vehicle (either dosed BID or QID). Subjects were given the Subject-Rated Ocular Pain Assessment to subjectively rate their pain.
  Higher scores were worse outcomes.
  The following scoring scale was used for ocular pain:
  0 = None
  1. Minimal
  2. Mild
  3. Moderate
  4. Moderately Severe
  5. Severe
Time Frame: Visit 6 (postoperative day 15)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% QID | KPI-121 1.0% BID | Vehicle of KPI-121
Number analyzed (Participants) | 127 | 124 | 124
score on a scale | 0.2 (0.50) | 0.2 (0.51) | 0.3 (0.73)
Statistical Analysis 1: Comparison: KPI-121 0.25% QID vs Vehicle of KPI-121; Test type: Superiority; p = 0.2589, ANCOVA; Mean Difference (Final Values) = -0.1 — Estimated value is the between-group difference on mean ocular pain score at Day 15
Statistical Analysis 2: Comparison: KPI-121 1.0% BID vs Vehicle of KPI-121; Test type: Superiority; p = 0.2132, ANCOVA; Mean Difference (Final Values) = -0.1 — Estimated value is the between-group difference in mean ocular pain score at Day 15

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time subjects signed the informed consent until they exited the study at the end of Visit 7 (up to Day 19).
Arm/Group | KPI-121 0.25% QID | KPI-121 1.0% BID | Vehicle of KPI-121
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/125 | 0/126
Serious Adverse Events (participants affected / at risk) | 2/129 | 1/125 | 2/126
Other Adverse Events (participants affected / at risk) | 13/129 | 6/125 | 20/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KPI-121 0.25% QID (N=129) | KPI-121 1.0% BID (N=125) | Vehicle of KPI-121 (N=126)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystoid macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KPI-121 0.25% QID (N=129) | KPI-121 1.0% BID (N=125) | Vehicle of KPI-121 (N=126)
eye pain (Eye disorders) | 2 (2) | 1 (1) | 5 (5)
photophobia (Eye disorders) | 3 (3) | 1 (1) | 3 (3)
punctate keratitis (Eye disorders) | 3 (3) | 1 (1) | 0 (0)
eye inflammation (Eye disorders) | 2 (2) | 0 (0) | 4 (4)
ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 5 (5)
headache (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
eye irritation (Eye disorders) | 1 (1) | 1 (1) | 3 (3)
corneal oedema (Eye disorders) | 2 (2) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreement between the Principal Investigator and the Sponsor restricts the PI's rights to discuss or publish trial results until after the first to occur of the following:

(a) publication of such multi-center clinical trial results; (b) notification by sponsor that such a multi-center clinical trial submission is no longer planned; or ( c) the eighteen ( 18) month anniversary of the completion, abandonment or termination of such multi-center clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT02163824/Prot_SAP_000.pdf